CLINICAL TRIAL: NCT06049732
Title: Psychometric Evaluation of the Electronic Pain Assessment Tool PainChek® Adult in Nursing Homes in the United States
Brief Title: PainChek® US Validation Nursing Home Study
Status: Completed | Type: Observational
Sponsor: PainChek Ltd (Industry)
Collaborators: Donawa Lifescience Consulting SRL (Unknown); TechnoSTAT Clinical Services (Unknown)
Responsible Party: Sponsor
Other Study IDs: PCK - US001/2020
Record Dates: First submitted 2023-09-10; First posted 2023-09-22 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Dementia; Pain
Keywords: Pain assessment
MeSH Terms: conditions — Dementia; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nursing home residents with moderate to severe dementia: Simultaneous pain assessments using PainChek® and the Abbey Pain Scale undertaken by two independent pain assessors, blinded to each others results
  Interventions: Device: PainChek®

INTERVENTIONS:
Device: PainChek® — Both PainChek® and the Abbey Pain Scale are observational pain assessment tools which have been designed to assist healthcare professionals and profession caregivers assess pain in people who cannot self-report their pain
  Other Names: Abbey Pain Scale

SUMMARY:
Pain is common amongst people living with dementia. However, as people's dementia worsens their ability to self-report pain diminishes because of limitations in their cognition and communication abilities. As a result pain in people with moderate to severe dementia often goes under-recognised and undertreated.

PainChek® is a technology-enabled, observational pain assessment tool, in the form of a mobile application designed specifically to assist healthcare professionals and professional caregivers assess pain in people with moderate severe dementia. In this study the investigators aim to assess the performance of PainChek® in assessing pain in nursing home residents with moderate to severe dementia compared to the Abbey Pain Scale.

DETAILED DESCRIPTION:
Study Design: This is a prospective, multicenter, observational study with the primary objective to validate PainChek® for assessing pain in subjects with moderate-to-severe dementia compared to the Abbey Pain Scale (APS).

In addition, the study data will be used to demonstrate test-retest reliability of the PainChek® device.

Study Objectives: PainChek® has been calibrated and successfully validated against the Abbey Pain Scale in Australia and the United Kingdom. The primary objective of the study is to demonstrate the validity of this calibration in the US intended use population.

As secondary objective, this study will the test-retest reliability of PainChek® as compared to the Abbey Pain Scale (APS).

As an additional exploratory objective, the association between respiratory rate (RR) and heart rate (HR) and pain scores detected by PainChek® and APS will be investigated.

Data generated in this study will be used in support of a United States Food and Drug Administration (FDA) De Novo submission.

Clinical Sites: The study will include between 5 and 12 nursing homes in the US.

Study Procedures: The study is entirely observational and follows the patient's standard of care (SOC).

Each participating site will assign raters providing pain assessments for the study. Each rater will be requested to assess pain of enrolled subjects using either the PainChek® device (PainChek® raters) or the Abbey Pain Scale (APS raters). Raters from all participating sites will be trained on the assessment tools by PainChek.

Consent to participate in the study will be requested from legally authorized representatives (LARs) of subjects with moderate-to-severe dementia potentially eligible to participate in the study. Following consent signature by the subject's LAR, subjects will be enrolled in the study. Weekly pain ratings of enrolled subjects will be done concurrently by two independent raters using PainChek® and the Abbey Pain Scale (APS). Pain assessments will be done twice (at rest and post movement) at each session. At the end of both the at rest and post movement pain assessments, the subject's respiratory rate (RR) and heart rate (HR) will be measured using a fingertip pulse oximeter. In addition, the study coordinator will document changes in clinical status of the resident between each encounter.

Raters will be blinded to each other's assessment, to prior pain assessments on the same subject and to subject's clinical status as assessed by the study coordinator. Each subject is planned to be assessed up to 10 times for maximum study duration per subject of 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled in the study should meet all of the following criteria:

  1. have been diagnosed with moderate-to-severe dementia on the basis of the score obtained with one of the following tools:

     1. Mini-Mental State Examination (MMSE) score < 19 OR
     2. MDS Cognitive Performance Scale (CPS) score > 3 OR
     3. Another cognitive assessment tool routinely used within the aged care facility allowing the identification of subjects with moderate-to-severe dementia
  2. are unable to reliably self-report pain as determined by the caregiver
  3. have been living in the aged care home for at least 30 days prior to the day of screening
  4. must have had an informed consent signed by the subject's legally authorized representative

Exclusion Criteria:

* Subjects enrolled in the study should not meet any of the following criteria:

  1. subject is unable to partially or completely exhibit any facial expression (e.g. as a result of a facial palsy, facial injuries or other pathologies)
  2. the treating physician determines it is inappropriate to assess the subject for pain
  3. subject is currently receiving or has received in the last 30 days prior to screening an investigational product and/or participated in another clinical trial.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include non-verbal subjects diagnosed with moderate to severe dementia living in nursing homes in the US. All comers will be evaluated for study eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
Change in pain score using PainChek Adult | Throughout the study on multiple occasions, on average every 7 days
  Change in pain measurement using PainChek Adult pain scale with the resident At Rest then Post Movement or vice versa. The scale includes 42 items across 6 domains, with scores of 0-6 representing No Pain, 7-11 Mild Pain, 12-15 Moderate Pain and 16-42 Severe Pain.
Change in pain score using Abbey Pain Scale | Throughout the study on multiple occasions, on average every 7 days
  Change in pain measurement using the Abbey Pain Scale with the resident At Rest then Post Movement or vice versa. The scale includes 18 items across 6 domains, with scores of 0-2 representing No Pain, 3-7 Mild Pain, 8-13 Moderate Pain and 14-18 Severe Pain.

OTHER OUTCOMES:
Change in heart rate using a finger pulse oximeter | Throughout the study on multiple occasions, on average every 7 days
  Change in heart rate measured using a Masimo MightySat™ Rx Finger Pulse Oximeter with the subject At Rest then Post Movement or vice versa
Change in respiratory rate using a finger pulse oximeter | Throughout the study on multiple occasions, on average every 7 days
  Change in respiratory rate measured using a Masimo MightySat™ Rx Finger Pulse Oximeter with the subject At Rest then Post Movement or vice versa

CONTACTS AND LOCATIONS:
Overall Officials: Kim Bergen-Jackson, PhD, Principal Investigator — Christian Retirement Services, Inc (Oaknoll); Wingyun Mak, PhD, Principal Investigator — The New Jewish Home
Locations (5):
- United States (5):
  - NewAldaya Lifescapes, Cedar Falls, Iowa
  - The Meth-Wick Community, Cedar Rapids, Iowa
  - Luther Manor Communities, Dubuque, Iowa
  - Oaknoll Retirement Residence, Iowa City, Iowa
  - The New Jewish Home, New York, New York

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Background] Atee M, Hoti K, Parsons R, Hughes JD. Pain Assessment in Dementia: Evaluation of a Point-of-Care Technological Solution. J Alzheimers Dis. 2017;60(1):137-150. doi: 10.3233/JAD-170375. PMID 28800333
- [Background] Atee M, Hoti K, Parsons R, Hughes JD. A novel pain assessment tool incorporating automated facial analysis: interrater reliability in advanced dementia. Clin Interv Aging. 2018 Jul 16;13:1245-1258. doi: 10.2147/CIA.S168024. eCollection 2018. PMID 30038491
- [Background] Hoti K, Atee M, Hughes JD. Clinimetric properties of the electronic Pain Assessment Tool (ePAT) for aged-care residents with moderate to severe dementia. J Pain Res. 2018 Jun 1;11:1037-1044. doi: 10.2147/JPR.S158793. eCollection 2018. PMID 29910632
- [Background] Atee M, Hoti K, Hughes JD. Psychometric Evaluation of the Electronic Pain Assessment Tool: An Innovative Instrument for Individuals with Moderate-to-Severe Dementia. Dement Geriatr Cogn Disord. 2017;44(5-6):256-267. doi: 10.1159/000485377. Epub 2018 Jan 23. PMID 29393207
- [Background] Babicova I, Cross A, Forman D, Hughes J, Hoti K. Evaluation of the Psychometric Properties of PainChek(R) in UK Aged Care Residents with advanced dementia. BMC Geriatr. 2021 May 28;21(1):337. doi: 10.1186/s12877-021-02280-0. PMID 34049501